CLINICAL TRIAL: NCT00215943
Title: Phase III Randomized Trial of Thalidomide/Dexamethasone vs VAD as Induction Chemotherapy for Newly Diagnosed Myeloma Patients and Evaluation of the Effects of Zoledronate on Chemotherapy Induced Apoptosis and Antigen Presentation.
Brief Title: Phase III Randomized Trial of Thalidomide/Dexamethasone Versus Vincristine+Adriamycin+Dexamethasone (VAD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor accrual, changes in management of newly diagnosed myeloma patients, new drugs/more effective regimens.
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13043; CZOL446E (Other: Novartis)
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Results first posted 2014-03-04 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2013-08

CONDITIONS: Multiple Myeloma
Keywords: hematologic malignancy
MeSH Terms: conditions — Multiple Myeloma; Hematologic Neoplasms | interventions — Zoledronic Acid; Dexamethasone; Calcium Dobesilate; Thalidomide; Vincristine; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VAD Treatment (Active Comparator): VAD (vincristine, adriamycin, dexamethasone). Vincristine and adriamycin was administered by continuous infusion via a venous catheter for 96 hours every 28 days. Each 28 days is considered one "cycle" of therapy. Patients were to receive 4 to 6 cycles of therapy. Dexamethasone was taken in pill form. During the first 2 cycles it was taken on days 1-4, 9-12, 17-20. For all other cycles dexamethasone was taken only on days 1-4. Patients were randomized to receive zoledronic acid IV on either Day 1 or 15 of each cycle.
  Interventions: Drug: zoledronic acid; Drug: vincristine; Drug: adriamycin
- Thalidomide and Dexamethasone Treatment (Active Comparator): Thalidomide was taken orally once every day in the evening for four to six months. The dexamethasone was taken in a pill form. During the first 2 cycles it was taken on days 1-4, 9-12, 17-20. For all other cycles dexamethasone was taken only on days 1-4.
  Interventions: Drug: zoledronic acid; Drug: dexamethasone; Drug: thalidomide

INTERVENTIONS:
Drug: zoledronic acid — Patients were randomized to receive zoledronic acid I.V. on either Day 1 or 15 of each cycle. This schedule continued monthly as long as the patient remained on study. The dose was calculated based on the patients' monthly creatinine clearance.
  Other Names: Zometa®; Zoledronate
Drug: dexamethasone — As outlined in VAD Treatment arm and Thalidomide and Dexamethasone Treatment arm
  Other Names: Decadron; NSC-34521
  Arms: Thalidomide and Dexamethasone Treatment
Drug: thalidomide — As outlined in Thalidomide and Dexamethasone Treatment arm
  Other Names: Thalomid™
  Arms: Thalidomide and Dexamethasone Treatment
Drug: vincristine — As outlined in VAD Treatment Arm
  Other Names: Oncovin; NSC-67574
  Arms: VAD Treatment
Drug: adriamycin — As outlined in VAD Treatment arm
  Other Names: Doxorubicin; NSC-123127
  Arms: VAD Treatment

SUMMARY:
Investigators planned to accrue 176 participants, to compare the response rate, overall response rate and survival of patients with multiple myeloma (MM) when randomized to two regimens (thalidomide+Dexamethasone versus Vincristine+Adriamycin+Dexamethasone). Investigators also planned to test if treatment with zoledronate immediately prior to chemotherapy results in an enhanced response to treatment (i.e. increase in complete response rates).

DETAILED DESCRIPTION:
Patients Randomized to receive VAD (vincristine, adriamycin, dexamethasone): All patients received four cycles of VAD repeated every 4 weeks. Chemotherapy was administered by continuous IV Infusion for 96 hours: vincristine at a dose of 0.4 mg/day and doxorubicin at a dose of 9 mg/m^2/day. Patients were administered dexamethasone 40 mg by mouth (PO) on days 1 to 4, 9 to 12, and 17 to 20 of the initial two cycles. Dexamethasone was given only on days 1-4 of all subsequent cycles. Patients were randomized to receive zoledronic acid IV on either Day 1 or 15 of each cycle. This schedule continued monthly as long as the patient remained on study. The dose was calculated based on the patients' monthly creatinine clearance. Upon initiation of Zometa therapy, the following guidelines were applied: For patients with creatinine clearance >60 mL/min, the recommended dose remained at 4mg. For patients with reduced creatinine clearance, dosing was calculated to achieve the same area under curve (AUC) as in patients with creatinine clearance of 75 mL/min. Creatinine clearance was calculated using the Cockcroft-Gault formula.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed MM confirmed by the presence of bone marrow plasmacytosis with > 10 percent plasma cells, sheets of plasma cells, or biopsy-proven plasmacytoma. Patients must have Durie-Salmon Stage IIA-B or IIIA-B. Patients with non-secretory myeloma are eligible. (These patients will not be included in the analysis of response rates, but will be assessed for toxicity and survival).
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, 2, or 3
* ≥ 18 years of age.
* Signed informed consent form
* Expected survival of greater than 8 weeks
* Capable of swallowing study medication tablets
* Capable of following directions regarding taking study medication, or has a daily care provider who will be responsible for administering study medication.
* Patients will be eligible for study even if they lack socioeconomic access to autologous transplantation. (These patients will be identified prior to randomization so as not to confound study results).
* All patients (in the event that they are randomized to the thalidomide/dexamethasone arm) must agree to take part in the "System for Education and Prescribing Safety" (S.T.E.P.S.)™. They must sign a separate informed consent for this program.

Exclusion Criteria:

* Elevated direct bilirubin > 2 mg/dl
* Serum alanine aminotransferase (ALT) or serum aspartate aminotransferase (AST) > 2 times the upper limit of normal (ULN)
* Absolute neutrophil count (ANC) <1000/mL, unless felt to be secondary to myeloma
* Ongoing radiation therapy, or radiation therapy within 3 weeks prior to first treatment, unless the acute side effects associated with such therapy are resolved.
* Prior treatment for multiple myeloma
* Prior bisphosphonate use is allowed but they must be discontinued before starting treatment.
* Concurrent uncontrolled serious infection
* Patients with peripheral (sensory) neuropathy, grade 3 or higher
* Life-threatening illness (unrelated to tumor)
* History of any other ACTIVE and INVASIVE cancer other than the present condition (except non-melanoma skin cancer), unless in complete remission and off of all therapy for that disease for a minimum of 3 years.
* Women of childbearing potential (unless utilizing birth control) or who are pregnant or nursing will be excluded from this study.
* Patients with comorbid conditions that would contraindicate the use of vincristine, doxorubicin, dexamethasone, thalidomide, or zoledronate.
* Plasma Cell Leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2003-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Alsina, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (5):
- United States (4):
  - Morton Plant Hospital, Clearwater, Florida
  - Watson Clinic, Lakeland, Florida
  - Fawcett Memorial Hospital, Port Charlotte, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
- San Juan VA Hospital, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began at Moffitt Cancer Center in June of 2003 and ended prematurely in December of 2007.
Pre-assignment Details: 90 participants were consented. 83 were eligible and randomized to treatment arms. 2 became ineligible after randomization and prior to treatment. 8 withdrew prior to treatment. 73 began treatment.
Groups:
- Active Comparator: VAD Treatment: VAD (vincristine, adriamycin, dexamethasone). Vincristine and adriamycin was administered by continuous infusion via a venous catheter for 96 hours every 28 days. Each 28 days is considered one "cycle" of therapy. Patients were to receive 4 to 6 cycles of therapy. Dexamethasone was taken in pill form. During the first 2 cycles it was taken on days 1-4, 9-12, 17-20. For all other cycles dexamethasone was taken only on days 1-4. Patients were randomized to receive zoledronic acid IV on either Day 1 or 15 of each cycle.
- Active Comparator: Thalidomide and Dexamethasone Treatment: Thalidomide was taken orally once every day in the evening for four to six months. The dexamethasone was taken in a pill form. During the first 2 cycles it was taken on days 1-4, 9-12, 17-20. For all other cycles dexamethasone was taken only on days 1-4.
Period: Overall Study
Arm/Group | Active Comparator: VAD Treatment | Active Comparator: Thalidomide and Dexamethasone Treatment
Started | 36 | 37
Completed | 27 | 23
Not Completed | 9 | 14
Not completed — Disease Progression | 3 | 5
Not completed — Alternate therapy | 0 | 1
Not completed — Adverse Event | 3 | 6
Not completed — Other disease | 0 | 1
Not completed — Other complications | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Comparator: VAD Treatment | Active Comparator: Thalidomide and Dexamethasone Treatment | Total
Number analyzed (Participants) | 36 | 37 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 27 | 52
  >=65 years | 11 | 10 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 21 | 23 | 44
Region of Enrollment [Number; unit: participants]
  United States | 36 | 37 | 73

OUTCOME MEASURES:

1. Primary Outcome: Response Rates of VAD vs. Thalidomide/Dexamethasone
Description: Blade (15) criteria for remission in multiple myeloma was used to assess response. Complete Response (CR)includes: Disappearance of the original monoclonal protein from the blood and urine on at least two determinations for a minimum of 6 weeks by immunofixation studies. Partial Response (PR) includes: At least a 50% reduction in the level of serum monoclonal protein for at least two determinations 6 weeks apart. Minimal Response (MR)includes: At least a 25% to 49% reduction in the level of serum monoclonal protein for at least 2 determinations 2 weeks apart.
Time Frame: End of Cycle 4 - 4 Months per Participant
Population: All evaluable participants
Measure: Number; unit: participants
Arm/Group | Active Comparator: VAD Treatment | Active Comparator: Thalidomide and Dexamethasone Treatment
Number analyzed (Participants) | 36 | 37
participants
  Complete Response | 1 | 1
  Partial Response | 9 | 16
  Minimal Response | 6 | 2

2. Secondary Outcome: Number of Participants With Adverse Events, by Group
Description: Number of participants with toxicities of Thalidomide/Dexamethasone vs. VAD as induction regimens in newly diagnosed multiple myeloma (MM).
Time Frame: 4 Years, 7 Months
Population: All evaluable participants
Measure: Number; unit: participants
Arm/Group | Active Comparator: VAD Treatment | Active Comparator: Thalidomide and Dexamethasone Treatment
Number analyzed (Participants) | 36 | 37
participants
  Serious Adverse Events (SAEs) | 0 | 1
  Adverse Events (AEs) | 36 | 37

3. Secondary Outcome: Number of Participants With Progression Free Survival (PFS), by Treatment Arm
Description: Number of participants with PFS for thalidomide/Dexamethasone vs. VAD with respect to progression free survival in newly diagnosed MM. Progressive Disease (PD): (for patients not in CR) Requires one or more of the following; > 25% increase in the level of serum monoclonal paraprotein, which must also be an absolute increase of at least 5 g/L and confirmed on a repeat investigation.
  > 25% increase in 24-hour urinary light chain excretion, which must also be an absolute increase of at least 200mg and confirmed on a repeat investigation.
  >25% increase in plasma cells in a bone marrow aspirate, which also must be an absolute increase of at least 10%. Definite increase in the size of existing lytic lesions or plasmacytomas. Development of new bone lesions or plasmacytomas (except compression fractures). Development of hypercalcemia (corrected calcium > 11.5 mg/dL not attributable to other causes).
Time Frame: 4 Months
Population: All evaluable participants
Measure: Number; unit: participants
Arm/Group | Active Comparator: VAD Treatment | Active Comparator: Thalidomide and Dexamethasone Treatment
Number analyzed (Participants) | 36 | 37
participants | 2 | 1

4. Secondary Outcome: Overall Survival (OS), by Treatment Arm
Description: Median OS for thalidomide/Dexamethasone participants vs. VAD participants. Months from On Study to Expired/Last Date Known Alive.
  Investigators had planned to accrue 176 participants to calculate median overall survival.
Time Frame: Up to 10 Years
Population: All participants with evaluable follow-up data.
Measure: Median (Full Range); unit: months
Arm/Group | Active Comparator: VAD Treatment | Active Comparator: Thalidomide and Dexamethasone Treatment
Number analyzed (Participants) | 26 | 20
months | 57 [0 to 114] | 56.5 [2 to 115]

ADVERSE EVENTS:
Time Frame: 5 years
Description: All participants who received treatment
Arm/Group | Active Comparator: VAD Treatment | Active Comparator: Thalidomide and Dexamethasone Treatment
Serious Adverse Events (participants affected / at risk) | 0/36 | 1/37
Other Adverse Events (participants affected / at risk) | 36/36 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator: VAD Treatment (N=36) | Active Comparator: Thalidomide and Dexamethasone Treatment (N=37)
Pneumonitis/pulmonary infiltrates - Grade 4 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary/Upper Respiratory - Other - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator: VAD Treatment (N=36) | Active Comparator: Thalidomide and Dexamethasone Treatment (N=37)
Abdominal pain or cramping (Gastrointestinal disorders) | 1 (1) | 2 (2)
Alkaline phosphatase (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 17 (18) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (4) | 7 (11)
Bilirubin (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 22 (27) | 23 (28)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 13 (15) | 24 (31)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Creatinine (Metabolism and nutrition disorders) | 7 (12) | 6 (14)
Dehydration (Gastrointestinal disorders) | 5 (7) | 6 (9)
Depressed level of consciousness (General disorders) | 0 (0) | 2 (2)
Diarrhea - patients without colostomy (Gastrointestinal disorders) | 4 (5) | 9 (10)
Dizziness/lightheadedness (General disorders) | 2 (3) | 6 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dyspepsia/heartburn (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 15 (17)
Dysuria (painful urination) (Renal and urinary disorders) | 0 (0) | 2 (2)
Edema (Blood and lymphatic system disorders) | 6 (7) | 12 (15)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 18 (20) | 17 (21)
Fever (in the absence of neutropenia) (General disorders) | 3 (3) | 6 (8)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 0 (0) | 2 (2)
Low Hemoglobin (Blood and lymphatic system disorders) | 34 (70) | 31 (81)
Hypercalcemia (Metabolism and nutrition disorders) | 5 (6) | 4 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (28) | 12 (23)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 4 (6)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypertension (Cardiac disorders) | 3 (3) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (4) | 2 (5)
Hypoalbuminemia (Blood and lymphatic system disorders) | 7 (8) | 7 (13)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (17) | 13 (19)
Hypokalemia (Metabolism and nutrition disorders) | 4 (10) | 5 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (6) | 2 (5)
Hyponatremia (Metabolism and nutrition disorders) | 7 (10) | 5 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 10 (15) | 11 (13)
Hypotension (Cardiac disorders) | 2 (3) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (2)
Infection without neutropenia (Infections and infestations) | 11 (14) | 10 (17)
Insomnia (General disorders) | 6 (6) | 6 (6)
Low Leukocytes (total WBC) (Blood and lymphatic system disorders) | 6 (11) | 7 (14)
Lymphopenia (Blood and lymphatic system disorders) | 5 (13) | 3 (12)
Melena/GI bleeding (Gastrointestinal disorders) | 1 (1) | 2 (2)
Mood alteration-anxiety, agitation (General disorders) | 3 (3) | 3 (3)
Mouth dryness (Gastrointestinal disorders) | 0 (0) | 2 (2)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (6)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 11 (15) | 8 (12)
Neuropathic pain (e.g., jaw pain, neurologic pain, phantom limb pain, post-infectious neuralgia, or (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neuropathy - motor (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (6)
Neuropathy - sensory (Musculoskeletal and connective tissue disorders) | 9 (9) | 14 (15)
Low Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 5 (9) | 6 (15)
Low Platelets (Blood and lymphatic system disorders) | 9 (20) | 10 (23)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (8)
Prothrombin time (PT) (Blood and lymphatic system disorders) | 0 (0) | 4 (11)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (8)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Rigors, chills (General disorders) | 2 (2) | 2 (2)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1) | 2 (5)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (2) | 3 (6)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 12 (12) | 3 (3)
Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 0 (0) | 2 (2)
Sweating (diaphoresis) (General disorders) | 2 (2) | 3 (3)
Syncope (fainting) (General disorders) | 0 (0) | 3 (3)
Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 3 (4) | 4 (4)
Thrombosis/embolism (Vascular disorders) | 7 (7) | 7 (7)
Transfusion - Platelets (Blood and lymphatic system disorders) | 2 (2) | 2 (4)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 6 (7) | 4 (8)
Tremor (General disorders) | 0 (0) | 7 (9)
Vomiting (Gastrointestinal disorders) | 2 (3) | 4 (5)
Weight loss (General disorders) | 3 (3) | 4 (5)

LIMITATIONS AND CAVEATS:
Target accrual for planned analysis (176) was not met. Principal Investigator (PI) determined study must close due to changes in the management of newly diagnosed myeloma (emergence of new drugs, more effective regimens).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes